CLINICAL TRIAL: NCT05124340
Title: Safety and Tuberculin Conversion Following BCG Vaccine Vial (Bio Farma) Compared to Registered BCG Vaccine (Bio Farma) in Indonesian Infants
Brief Title: Safety and Tuberculin Conversion Following BCG Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BS BCG 0221
Record Dates: First submitted 2021-10-26; First posted 2021-11-17 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: BCG Vaccination Reaction
Keywords: BCG Vaccine; Safety of BCG Vaccine; Tuberculin Conversion

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Observer Blind : Investigational Product and Active Comparator are masking. Lot number is masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): 1 dose of BCG vial vaccine injected in right deltoid armintradermally
  Interventions: Biological: BCG vial vaccine
- Active Comparator (Active Comparator): 1 dose of BCG ampoule vaccine injected in right deltoid arm intradermally
  Interventions: Biological: BCG ampoule vaccine

INTERVENTIONS:
Biological: BCG vial vaccine — Intradermal injection
  Arms: Vaccine
Biological: BCG ampoule vaccine — Intradermal injection
  Arms: Active Comparator

SUMMARY:
The study is an bridging study, observer-blind, randomized, controlled prospective intervention study. The primary objective is evaluate the safety of BCG Vaccine Vial (Bio Farma).

DETAILED DESCRIPTION:
This trial is bridging study, observer blinded, comparative, randomized study. Approximately 220 subjects will be recruited, 110 subjects are the investigational arm and 110 subjects are the active comparator arm.

The objective of the study is to evaluate the safety of BCG Vaccine Vial (Bio Farma), and assess the the local and systemic reactions within 90 days after vaccination in each group, and assess the tuberculin conversion in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infant aged 0-1 month.
2. Infants born after 37-42 weeks of pregnancy.
3. Infant weighing 2500 gram or more at birth.
4. Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.
5. Parents will commit themselves to comply with the instructions of the investigator and with the schedule of the trial.

Exclusion Criteria:

1. Child concomitantly enrolled or scheduled to be enrolled in another trial.
2. Evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature 37.5 celcius degrees).
3. Suspected of allergy to any component of the vaccines.
4. Newborn suspected of congenital or acquired immunodeficiency.
5. Received or plans to receive any treatment likely to alter the immune response intravenous (immunoglobulins, blood-derived products or long term corticotherapy (> 2 weeks)).
6. Received other vaccination with the exception of OPV and Hepatitis B vaccine.
7. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
8. Any skin disease such eczema generalisata other skin infection which makes difficult the assessment of the local reactios.
9. Mothers with HbsAg and HIV positive (by rapid test)
10. Parents planning to move from the study area before the end of study period.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of BCG Vaccine Vial (Bio Farma) | 30 minutes after vaccination
  Number and percentage of subject experience local reactions and systemic events occurring within 30 minutes after vaccination.

SECONDARY OUTCOMES:
To assess the local and systemic reactions within 30 minutes, 24 hours, 48 hours, 72 hours, 7 days and 30 days after vaccination. | 30 days after vaccination
  Number and percentage of subject experience ;ocal reactions and systemic events occurring within 24 hours, 48 hours, 72 hours, 7 days and 30 days after vaccination will be assessed per group with 95% CI.
To assess local reactions at 60 days and 90 days after vaccination in each group. | 90 days after vaccination
  Number and percentage of subject experience local reactions at 60 days and 90 days after vaccination will be assessed per group with 95% CI.
To assess serious adverse events within 30 days after vaccinantion in each group. | 30 days
  Number and percentage of subject experience Serious Adverse Events within 30 days after vaccination will be described.
To assess the tuberculin conversion in each group. | 2 days
  Number and percentage of subject who have tuberculin conversion

CONTACTS AND LOCATIONS:
Overall Officials: Dominicus Husada, MD, Principal Investigator — RS DR Soetomo Surabaya
Locations (1):
- Puskesmas Cerme, Gresik, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No